CLINICAL TRIAL: NCT01601158
Title: Safety and Efficacy of Allogeneic Umbilical Cord Blood Therapy for Children With Global Developmental Delay
Brief Title: Umbilical Cord Blood Therapy for Children With Global Developmental Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MinYoung Kim, M.D. (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, M.D., Associate Professor, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDDUCB
Record Dates: First submitted 2012-05-16; First posted 2012-05-17 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Global Developmental Delay
Keywords: Global developmental delay; Umbilical cord blood; Rehabilitation
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Umbilical Cord Blood and Rehabilitation (Experimental): Allogeneic Umbilical Cord Blood infusion and Active Rehabilitation
  Interventions: Biological: Umbilical Cord Blood administration; Other: Active Rehabilitation

INTERVENTIONS:
Biological: Umbilical Cord Blood administration — The subjects will be undertaken allogeneic umbilical cord blood infusion intravenously or intraarterially under non-myeloablative immunosuppression.
  Other Names: Donated Umbilical Cord Blood Units from Affiliated Cord Blood Bank
Other: Active Rehabilitation — All subjects should participate in active rehabilitation. They will receive two physical and occupational therapy sessions per day. Post discharge, each participant should continue to receive rehabilitation therapy at least 3 days per week until the study completion.

SUMMARY:
This open-label study aims to evaluate the safety and efficacy of umbilical cord blood therapy for children with global developmental delay.

DETAILED DESCRIPTION:
Global developmental delay (GDD) is a subset of developmental disabilities defined as significant delay in two or more of the following developmental domains: gross/fine motor, speech/language, cognition, social/personal, and activities of daily living.

Umbilical cord blood has been used for inherited metabolic diseases that feature global developmental delay and many experimental animal studies have revealed umbilical cord blood is useful to repair neurological impairments in brain.

ELIGIBILITY:
Inclusion Criteria:

* Global developmental delay
* Willing to comply with all study procedure

Exclusion Criteria:

* Medical instability including pneumonia or renal function at enrollment
* Poor cooperation of guardian,including inactive attitude for rehabilitation and visits for follow-up
* Uncontrolled persistent epilepsy
* Not eligible according to the principal investigator

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in Cognition | Baseline - 6 months - 12 months
  Korean Wechsler Preschool and Primay Scale of Intelligence (K-WPPSI) (Higher value means better cognitive function (K-WPPSI: below 70 - worst, over 130 - best). The investigators will report K-WPPSI at each assessment time points.
Changes in Cognitive Neurodevelopmental Outcome | Baseline - 1 month - 3 months - 6 months - 12 months
  Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Mental Scales (Higher value means better cognitive function, K-BSID-II mental scale raw score: 0 - worst, 178 - best). The investigators will report K-BSID-II Mental Scale raw scores at each assessment time points.

SECONDARY OUTCOMES:
Changes in Motor Performance | Baseline - 1 month - 3 months - 6 months - 12 months
  GMPM (Gross Motor Performance Measure) as a standardized measurement tool for assessing quality of movement regarding 3 properties of 5 ones; alignment, coordination, dissociated movement, stability, and weight shift (range: 0~100, Higher value means better motor quality). The investigators will report GMPM scores at each assessment time points.
Changes in Standardized Gross Motor Function | Baseline - 1 month - 3 months - 6 months - 12 months
  GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 , Higher value means better gross motor function). The investigators will report GMFM scores at each assessment time points.
Changes in Motor Neurodevelopmental Outcome | Baseline - 1 month - 3 months - 6 months - 12 months
  Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Motor Scales (higher value means better motor function: 0 - worst, 111 - best). The investigators will report K-BSID-II Motor Scale raw scores at each assessment time points.
Changes in Functional Independence in Daily Activities | Baseline - 1 month - 3 months - 6 months - 12 months
  WeeFIM (Functional Independence Measure for Children) measures functional independence in daily activities. WeeFIM contains 18 items and each item is ranked from complete dependence (scored as 1) to complete independence (scored as 7). The range is from 18 to 126 and higher scores mean more independent performance in daily activities. The investigators will report total WeeFIM scores measured at each assessment time points.
Changes in Visual Perception Test | Baseline - 1 month - 3 months - 6 months - 12 months
  We will evaluate visual perception function with one of three measures: DTVP (Developmental Test of Visual Perception), MVPT (Motor-free Visual Perception Test), and VMI (Visual-Motor Integration, Visual Perception and Motor Coordination). All can be scored as percentile rank from 0 to 100. Higher values mean better visual perception ability
Changes in Muscle Strength | Baseline - 1 month - 3 months - 6 months - 12 months
  Summation of MMT (manual muscle strength test score): summated scores of the manual muscle strength test (zero=0, trace=1, poor=2, fair=3, good=4, normal=5) for flexors, extensors, abductors, and adductors of bilateral shoulder and hip joints; flexors and extensors of bilateral elbow, wrist, and knee; dorsiflexors and plantar flexors of the ankles (range: 0 ~ 160) Higher scores mean better muscle strength. Categories of outcome table will be summation of MMT scores measured at each assessment time point.
Changes in Functional Performance in Daily Activities | Baseline - 1 month - 3 months - 6 months - 12 months
  Pediatric Evaluation of Disability Inventory (PEDI) for assessing functional performance in daily activities in children (All values are adjusted and higher value means better functional performance, 0 - worst, 100 - best). We will report 2 scales and 3 domains of each scale: a Functional Skill Scale (FSS) and a Caregiver Assistance Scale (CAS) which are divided respectively into 3 domains: self care, mobility, and social function. Categories of outcome table will be each domain scores measured at each assessment time point.
Changes in Language Evaluation | Baseline - 6 months - 12 months
  Sequenced Language Scale for Infant (SELSI), Preschool Receptive-Expressive Language Scale (PRES) or Korean Western Aphasia Battery (K-WAB) will be used depending on age and function.

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea